CLINICAL TRIAL: NCT02986100
Title: An Open-Label, Non-Randomized, Phase I Study to Assess the Absorption, Metabolism, and Excretion Following a Single Oral Dose of [14C]-Rucaparib in Patients With Advanced Solid Tumors
Brief Title: Absorption, Metabolism, and Excretion Following a Single Oral Dose of [14C]-Rucaparib
Acronym: AME
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: pharmaand GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CO-338-045; 2015-004394-32 (EudraCT Number)
Record Dates: First submitted 2016-11-14; First posted 2016-12-08 (Estimated); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Solid Tumor
Keywords: rucaparib; CO-338; Clovis; Clovis Oncology; PARP inhibitor; Absorption; Metabolism; Excretion
MeSH Terms: interventions — rucaparib

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (1):
- C-14 labeled rucaparib (Experimental): Each patient will receive a single oral dose of 600 mg [14C] rucaparib (approximately 140 µCi) in the fasted state. Patients will be confined at the study site for the collection of blood samples and excreta for a maximum of 13 days, from Day -1. The patient can be discharged sooner than Day 13, if the discharge criteria are met.
  After completion of Part I, patients with a deleterious BRCA mutation will have the option to participate in Part II by receiving 600 mg BID rucaparib tablets orally in 28 day cycles until disease progression, unacceptable toxicity, death, or discontinuation for other reasons
  Interventions: Drug: C-14 labeled Rucaparib; Drug: Rucaparib

INTERVENTIONS:
Drug: C-14 labeled Rucaparib — Each dosage unit consists of a hard gelatin capsule filled with cold rucaparib camsylate and [14C]-rucaparib camsylate salt. Each capsule contains approximately 150 mg rucaparib (free base weight) and approximately 35 µCi of [14C]-rucaparib. Each patient will ingest four capsules in the fasted state for a total dose of 600 mg rucaparib (free base weight) with approximately 140 µCi of [14C]-rucaparib
Drug: Rucaparib — 200 & 300 mg tablet
  Other Names: CO-338; Rubraca

SUMMARY:
The purpose of this study is to characterize the mass balance, absorption, metabolism, and elimination pathways of orally administered [14C] rucaparib followed by cycle by cycle treatment with rucaparib continuing until disease progression or other reason for discontinuation

DETAILED DESCRIPTION:
This is a Phase 1, open-label, non-randomized, mass balance study in patients with histologically or cytologically confirmed advanced solid tumors. Approximately 6 patients will be enrolled. The study will consist of 2 parts: a mass balance part (Part I) and a rucaparib treatment part (Part II).

Each patient will receive a single oral dose of 600 mg [14C] rucaparib (approximately 140 µCi) in the fasted state. Patients will be confined at the study site for the collection of blood samples and excreta for a maximum of 13 days, from Day -1. The patient can be discharged sooner than Day 13, if the discharge criteria are met. If the cumulative recovery of radioactivity exceeds 90% of the administered dose or if radioactivity in urine and feces is < 1% of the administered dose over a 24 hour period on two consecutive days, as determined by quick counts.

In Part II, the treatment with rucaparib in 28-day cycles will continue until progression of disease, unacceptable toxicity, or other reason for discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced solid tumor
* Part II only: Have a known deleterious BRCA1/2 mutation (germline or somatic) as determined by a local or central laboratory
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate bone marrow, renal, and liver function

Exclusion Criteria:

* Prior treatment with chemotherapy, radiation, antibody therapy or other immunotherapy, gene therapy, vaccine therapy, or angiogenesis inhibitors within 14 days prior to Day 1
* Participation in a trial involving administration of [14C]-labeled compound(s) within the last 6 months prior to Day 1
* Arterial or venous thrombi (including cerebrovascular accident), myocardial infarction, admission for unstable angina, cardiac angioplasty, or stenting within the last 3 months prior to Screening
* Pre-existing duodenal stent, recent or existing bowel obstruction, and/or any gastrointestinal disorder or defect that would, in the opinion of the Investigator, interfere with absorption of rucaparib
* Untreated or symptomatic central nervous system (CNS) metastases
* Evidence or history of bleeding disorder
* Participation in another investigational drug trial within 14 days prior to Day 1 (or 5 times the half-life of the drug, whichever is longer) or exposure to more than three new investigational agents within 12 months prior to Day 1
* Acute illness (eg, nausea, vomiting, fever, diarrhea) within 14 days prior to Day 1, unless mild in severity and approved by the Investigator and Sponsor's/designated medical representative
* Active second malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of 14C-labeled rucaparib (radioactivity in whole blood and plasma): tmax | Days 1-13
  Time to peak concentration (tmax)
Pharmacokinetics of 14C-labeled rucaparib(Radioactivity in whole blood and plasma): Cmax | Days 1-13
  peak (maximum) concentration (Cmax)
Pharmacokinetics of 14C-labeled rucaparib(Radioactivity in whole blood and plasma): t1/2 | Days 1-13
  Elimination half-life (t1/2)
Pharmacokinetics of 14C-labeled rucaparib(Radioactivity in whole blood and plasma): AUC | Days 1-13
  Area under curve (AUC)
Pharmacokinetics of 14C-labeled rucaparib(Radioactivity in whole blood and plasma): CL/F | Days 1-13
  Oral clearance (CL/F)
Pharmacokinetics of 14C-labeled rucaparib(Radioactivity in whole blood and plasma): V/F | Days 1-13
  Apparent volume of distribution (V/F)
Excretion rate of 14C-labeled rucaparib(radioactivity in feces) | Days 1-13
  Percent of dose excreted in feces
Excretion rate of 14C-labeled rucaparib(radioactivity in urine) | Days 1-13
  Percent of dose excreted in urine
Pharmacokinetics of rucaparib (in urine): CLR | Days 1-13
  Renal clearance (CLR)
Excretion rate of 14C-labeled rucaparib(radioactivity in vomit, if applicable) | Days 1-13
  Percent of dose in vomit, if applicable
Metabolite identification of rucaparib in plasma, urine and feces | Days 1-13
Cumulative whole blood:plasma ratio calculated for Cmax | Days 1-13
  peak concentration (Cmax)
Cumulative whole blood:plasma ratio calculated for AUC0-tlast | Day 1-13
  AUC from time zero to the last time point with concentration above the lower limit of quantitation (AUC0-last)
Cumulative whole blood:plasma ratio calculated for AUCinf | Day 1-13
  AUC from time zero to infinity (AUCinf)

SECONDARY OUTCOMES:
Tolerability and safety of rucaparib assessed by incidence of Adverse Events (AEs), clinical laboratory abnormalities, and dose modifications | From cycle 1 Day 1 until radiologically confirmed disease progression, death, or initiation of subsequent treatment whichever comes first up to 52 weeks
  Incidence of Adverse Events (AEs), clinical laboratory abnormalities, and dose modifications

OTHER OUTCOMES:
To evaluate the antitumor activity of rucaparib in BRCA mutated solid tumors based on Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Cycle 1 Day 1 until progression of disease, unacceptable toxicity, or discontinuation for other reasons
  Response will be determined using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 and tumor markers per applicable criteria for a given tumor type

CONTACTS AND LOCATIONS:
Locations (1):
- PRA Magyarország Kft., Budapest, Rottenbiller Utca 13, Hungary

IPD SHARING:
Plan to Share IPD: No